CLINICAL TRIAL: NCT01311167
Title: Prospective Randomized Double Blind Placebo Controlled Intervention Study of the Effect of Dexamethasone on the Sodium Retention in Patients With Liver Cirrhosis
Brief Title: Treatment of Sodium Retention in Liver Cirrhosis With Dexamethasone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment problems (not enough patients were found who met eligibility criteria)
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Geneva (Other); University of Lausanne Hospitals (Other)
Responsible Party: National Center of Competence Kidney.CH, Swiss National Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dexa_Cirr_2011
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Liver Cirrhosis
Keywords: Dexamethasone; Sodium
MeSH Terms: conditions — Liver Cirrhosis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Daily administration of 2 mg of dexamethasone for 4 days
  Arms: Dexamethasone
Drug: Placebo — Daily administration of 2 mg of placebo for 4 days
  Arms: Placebo

SUMMARY:
Accumulation of salt and water in patients with liver disease (so called liver cirrhosis) is possibly related to the increased effect of steroid hormones on salt reabsorption in the kidney. By reducing overall steroid production with the dexamethasone the accumulation of salt and water could be prevented.

ELIGIBILITY:
Inclusion Criteria:

* patients with established liver cirrhosis (biopsy or biochemically)
* hepatorenal syndrome type 1 or 2 (with a serum creatinin >175 umol/l)
* age between 18 and 75
* no bacterial infection
* no cardiovascular or extrahepatic disease (end of life)
* no structural kidney disease
* no hepatocellular carcinoma

Exclusion Criteria:

* age under 15 or over 75
* treatment with corticosteroids (dexamethasone included)
* bacterial infection
* cardiovascular or extrahepatic disease (end of life)
* structural kidney disease (indicated by hematuria, proteinuria)
* hepatocellular carcinoma
* mental disability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Daily sodium excretion of sodium in the urine | 4 days

SECONDARY OUTCOMES:
Daily potassium excretion | 4 days
weight reduction | 4 days
Reduction of doses of diuretics | 4 days
Reduction of ascites | 4 days
Reduction of cortisol excretion in the urine | 4 days
Reduction of cortisol levels in the urine | 4 days

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - University Hospital Inselspital, Bern, Canton of Bern
  - University Hospital Geneva, Geneva, Canton of Geneva
  - University Hospital Lausanne, Lausanne, Canton of Vaud